CLINICAL TRIAL: NCT04234815
Title: Evaluating Impacts of a Brief Psychosocial Workshop for Veterans and Their Families in Ukraine
Brief Title: Evaluating Impacts of CSS for Veterans and Their Families in Ukraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9782
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Psychosocial Problem; Psychological Distress; Engagement, Patient
Keywords: Mental health; Psychosocial support; Intervention; Depression; Post-traumatic stress; Functioning
MeSH Terms: conditions — Patient Participation; Psychological Well-Being; Depression | interventions — Safety

STUDY DESIGN:
Masking Description: Participants are not informed of their condition, but may reasonably deduce it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CETA Short Session (CSS) (Experimental): A single-session, 1.5-2 hour group workshop that includes psychoeducation, self-assessment, safety screening, and training in cognitive coping. Participants with at least moderate symptoms of distress will also receive a follow-up phone call to discuss next steps occurring within one week after workshop attendance. On this phone call they will also be asked about their use of the cognitive coping skill over the last week, and provided feedback if using it incorrectly.
  Interventions: Behavioral: CETA Short Session (CSS)
- Enhanced Treatment as Usual (eTAU) (Active Comparator): A single-session, approximately 1-hour group workshop that includes the same psychoeducation, self-assessment, and safety screening as the experimental condition, but no training in cognitive coping. Participants with at least moderate symptoms of distress will also receive a follow-up phone call to discuss next steps occurring within one week after workshop attendance.
  Interventions: Behavioral: Psychoeducation and Safety

INTERVENTIONS:
Behavioral: CETA Short Session (CSS) — CETA Short Session (CSS) is a brief, low-intensity psychosocial intervention incorporating foundational components of the Common Elements Treatment Approach (CETA). CETA is an 8-12 session, transdiagnostic psychotherapy for common mental disorders. CSS was designed to serve as both a prevention/support approach for a broader range of needs, as well as an engagement/outreach strategy to identify and refer individuals to treatment. CSS is delivered in a group format over approximately two hours and consists of: 1) Psychoeducation: instruction about the brain and brain functioning, including normalization of psychological responses to stress and a brief self-assessment; 2) Safety: screening and referral for individuals identified as at risk of harm to self or others; and 3) Cognitive coping: based on the cognitive triangle, participants practice identifying an unhelpful thought changing it to a more helpful alternative, and examining how these thoughts impact feelings and behaviors.
  Arms: CETA Short Session (CSS)
Behavioral: Psychoeducation and Safety — This intervention is the same as CSS with the exception that the cognitive coping skill training is removed.
  Arms: Enhanced Treatment as Usual (eTAU)

SUMMARY:
This cluster-randomized controlled trial (c-RCT) evaluates the effectiveness of a brief, single-session psychosocial workshop, "CETA Short Session" (CSS), for reducing symptoms of distress and functional impairment and increasing treatment engagement among conflict veterans and their families in Ukraine. The CSS workshop includes psychoeducation, review of a self-assessment, safety screening, and training in cognitive coping. This will be evaluated against a single-session comparison workshop that includes all of the same workshop elements except for cognitive coping. Registration for both conditions includes completion of a self-assessment. Participants with safety concerns or very severe symptoms will be immediately referred to mental health treatment; others will be asked to wait for one month before being reassessed and, if indicated, referred to mental health treatment. Both conditions include an individual check-in phone call one week after the workshop. Distress and functional impairment outcomes will be assessed one month from baseline. Treatment engagement outcomes will be assessed three months from referral. The investigators hypothesize that individuals attending sessions randomized to CSS will show greater improvement in mental health outcomes and greater treatment engagement than those attending sessions randomized to the comparison condition.

With the onset of the COVID-19 pandemic in Spring 2019, the RCT was paused to develop and pilot an online version of both the CSS and comparison workshop. The trial protocol has now been expanded to continue the effectiveness trial while allowing for both online and [when/if feasible] in-person intervention delivery.

DETAILED DESCRIPTION:
Community-based organizations in Ukraine that are currently providing social services to veterans or their families and are interested in receiving training to provide CSS will be engaged as implementing partners. Individuals selected to be providers at these organizations will complete a 2-day Provider Training and will additionally receive ongoing supervision over the course of the study to ensure intervention fidelity and appropriate response and support to individuals needing referral to mental health treatment.

Cluster-level randomization to CSS or eTAU will be carried out at the workshop level within provider, such that all Providers will deliver both the CSS and eTAU workshops to groups that have been randomly allocated to either receive CSS or eTAU. In this way, all organizations will offer both CSS and eTAU, integrated into each organization's regular program offerings and advertised through organizations' regular communication channels.

As part of the registration and triage procedures included as regular programming in both arms of the trial, participants will self-complete a short, locally validated Self-Assessment Form that assesses symptoms of distress (depression, post-traumatic stress), functional impairment, and safety risk (two safety-related questions assessing recent thoughts of harm to self or others). This assessment will be completed in advance and reviewed by an M&E staff member prior to the workshop, but assessment scores will not determine workshop eligibility (e.g., people with low scores can still participate). One exception to this is that any individuals who respond positively to either of the safety questions will be contacted by the CSS/eTAU provider within 24-hours for further safety assessment. If no safety issues are identified, they will be registered for the workshop as normal; however, identified safety issues will trigger an appropriate safety planning or referral response as described below, which may include bypassing the workshop in lieu of direct enrollment in treatment services. At the end of the workshop, participants will be informed of the study and invited to participate; those who agree will provide informed consent.

After the workshop, as part of regular programming the provider will follow up individually with participants to discuss recommended next steps. Evaluation of level of need, and therefore choice of follow-up response, will be made by the provider using the self-assessment results as well as any information reported to the provider during the workshop (such as new safety concerns, or changes in problem scores). Follow-up contacts will be ordered by priority.

1. Individuals who indicate any new safety concerns at the workshop will be contacted within 24 hours for further assessment to determine the appropriate referrals and/or safety plan.
2. Individuals with high symptom scores, but no safety concerns, will be contacted within 72 hours and offered a referral to outpatient mental health care.
3. Individuals with moderate symptom scores will be contacted within 1 week for triage and encouraged to use the newly learned skills over the next month. On that triage phone call, participants will be told they will be re-assessed in one month to determine if they still require mental health treatment (at which time they would be referred if indicated). For those who attended CSS (rather than eTAU), providers will also ask about participant use of the cognitive coping skill over the past week, including asking them how often they've used it, whether it has been helpful, and soliciting an example through a series of questions that walk them through the skill.

At one month, all study participants who were not immediately referred to outpatient mental health services at baseline will be sent an individual link to re-administer the self-assessment, the CSS skill check, and complete an implementation feedback questionnaire.

For all study participants who receive an outpatient mental health referral, either immediate or delayed, engagement outcomes will be assessed three months following referral.

ELIGIBILITY:
Inclusion Criteria:

* Ukrainian adults (age 18 or older) who are Veterans of the Anti-Terrorist Operations (ATO) in Ukraine or an adult family member of a veteran
* Meets a minimum total problem score on the locally validated screener indicative of at least moderate symptoms of distress

Exclusion Criteria:

* People who identify as ATO veterans but are still active (i.e., active duty) in the Ukrainian military.
* Participants who arrive late to the workshop, operationalized as not having time to participate in the self-assessment review, will be excluded. In online workshops, late-arriving participants will be redirected to a waiting room, where they will be encouraged to attend a future session instead (and if so, could be included in the study). For in-person workshops, due to travel and other efforts required for attendance late arriving participants will be allowed to join the workshop, but excluded from the study due to lacking sufficient exposure. They can also choose to attend a future workshop, but if attending a portion of an initial workshop would remain study ineligible because they could potentially be exposed to both arms of the study.
* Participants who are identified by service providers as needing higher-level care rather than outpatient psychotherapy will be immediately referred to that care and excluded from the study. This exclusion criteria refers to imminent danger to self or others that requires urgent safety procedures and institution-based mental health care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1193 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Change in mental health symptom scores | Baseline, 1-month follow-up
  International Depression Symptom Scale (IDSS): a locally-validated self-report instrument that produces total and syndrome-specific scores. (range: 0-54, higher indicates more symptomatic)
Mental health treatment engagement | 3 months following referral to mental health treatment
  Follow-up on referral to mental health treatment, derived from client monitoring records (indicated as yes/no)
Change in functional impairment | Baseline, 1-month follow-up
  a locally developed (based on qualitative data) and validated self-report instrument that produces a functional impairment score (range: 0-56, higher scores indicate greater functional impairment)

SECONDARY OUTCOMES:
Aggression | Baseline, 1-month follow-up
  Items adapted (based on qualitative data) from the Conflict Tactics Scale - Revised (range: 0-18, higher scores indicate more aggression)
Social Connectedness | Baseline, 1-month follow-up
  Items adapted (based on qualitative data) from the Social Connectedness Scale - Revised (range: 0-24, higher scores indicate greater disconnection)
Alcohol consumption | Baseline, 1-month follow-up
  AUDIT-C scores (range: 0-12, higher scores indicate greater substance use)

OTHER OUTCOMES:
Implementation outcomes | 1-month follow-up
  JHU Implementation Measure for LMIC (JHUIM): A validated implementation questionnaire assessing adoption, acceptability, appropriateness, and feasibility of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Bass, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- NaUKMA, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No